CLINICAL TRIAL: NCT06052293
Title: A Phase 1 Open-Label, Multicenter Study to Assess the Safety and Efficacy of ANG003 in Patients With Exocrine Pancreatic Insufficiency Due to Cystic Fibrosis
Brief Title: Phase 1 Study to Assess Safety and Efficacy of ANG003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anagram Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANG003-22-101
Record Dates: First submitted 2023-08-09; First posted 2023-09-25 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Exocrine Pancreatic Insufficiency
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ANG003 Dose Level 1 (Experimental): Single administration starting dose contains lipase, protease and amylase.
  Interventions: Drug: ANG003
- ANG003 Dose Level 2 (Experimental): Single administration dose contains 2x lipase, 2x protease and 2x amylase starting dose.
  Interventions: Drug: ANG003
- ANG003 Dose Level 3 (Experimental): Single administration dose contains 4x lipase, 2x protease and 2x amylase starting dose.
  Interventions: Drug: ANG003
- ANG003 Dose Level 4 (Experimental): Single administration dose contains 6x lipase, 3x protease and 3x amylase starting dose.
  Interventions: Drug: ANG003

INTERVENTIONS:
Drug: ANG003 — To evaluate four possible combinations of lipase, protease and amylase.
  Other Names: Dose Level 1, Dose Level 2, Dose Level 3, and Dose Level 4.

SUMMARY:
Randomized, parallel, active-treatment Phase 1 study of a single dose of orally administered ANG003 with a test meal in adult subjects with cystic fibrosis-related exocrine pancreatic insufficiency. The study's overall objectives are to evaluate the safety, tolerability and effect of four dose levels of ANG003.

DETAILED DESCRIPTION:
The Phase 1 study was designed to compare a 24h Baseline Substrate Absorption Challenge Test (SACT) period with no enzymes to a 24h ANG003 SACT period with enzymes. Eligible subjects will be randomly assigned with equal allocation to one of four active dose levels of lipase, protease and amylase. Approximately 48 to 60 eligible subjects are planned to be enrolled in the study with 12 to 15 subjects assigned to each dose level from up to 21 investigational sites.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years of age or older.
2. Confirmed diagnosis of CF defined as: a) CF signs and symptoms AND b) Two CF-causing mutations on genetic testing or sweat chloride >60 mEq/L.
3. Documented history of fecal elastase <100 µg/g stool.
4. EPI clinically controlled with minimal clinical symptoms and on a stable dose of PERT for 90 days before screening as determined by the Investigator.
5. Adequate nutritional status measured by body mass index ≥20kg/m2 for adult subjects.

Exclusion Criteria:

1. Subjects with diabetes mellitus who are unable to refrain from short-acting and rapid-acting insulin on Days 1 and 5 for a daily total of 6 hours.
2. Involuntary loss of ≥10% of usual body weight within last 6 months or involuntary loss of >5% of body weight within 1 month.
3. Requires use of naso-gastric, J-tube, G-tube, and/or enteral feeding for the study duration.
4. CF pulmonary exacerbation within 30 days prior to the Baseline SACT Period (Visit 2).
5. Subjects who cannot discontinue omega-3 supplements >500 mg of DHA and EPA daily.
6. Subjects unable to tolerate missing a dose of PERT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE), Serious Adverse Events (SAE), and AEs Leading to Study Discontinuation | Assessed through study completion, up to 9 days (Day 1 thru Day 9).
  AE, SAE, and AEs leading to study discontinuation measured by frequency and severity during study.
Malabsorption Symptoms | Acute PAGI-SYM is based upon 7-day recall.
  Severity of malabsorption symptoms (e.g., abdominal discomfort or pain, bloating, heartburn, regurgitation or reflux, retching, stomach fullness, and vomiting) by patient reported outcome scale (0=None; 1=Very Mild; 2=Mild; 3=Moderate; 4=Severe; 5=Very Severe). Measured by 20 questions contained in Acute Patient Assessment of Gastrointestinal Symptoms (Acute PAGI-SYM) questionnaire.

SECONDARY OUTCOMES:
Fat Absorption | Assessed through study completion, up to 9 days (Day 1 thru Day 9).
  Measured by concentration and percent of plasma fatty acids.
Protein Absorption | Assessed through study completion, up to 9 days (Day 1 thru Day 9).
  Measured by changes in plasma concentration of amino acids.
Carbohydrate Absorption | Assessed through study completion, up to 9 days (Day 1 thru Day 9).
  Changes in glucose (mg/dL) as measured by continuous glucose monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Meghana Sathe, MD, Principal Investigator — University of Texas
Locations (20):
- United States (20):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Long Beach Memorial Medical Center, Long Beach, California
  - National Jewish Health, Denver, Colorado
  - Norton Children's Research Institute affiliated with University of Louisville School of Medicine, Louisville, Kentucky
  - Massachusetts General Hospital,, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Harper University Hospital / Wayne State University, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical College, Albany, New York
  - New York Medical College at Westchester Medical Center, Valhalla, New York
  - Akron Childrens Hospital, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No